CLINICAL TRIAL: NCT06749483
Title: The Gut Microbiome - Source of Sepsis and Novel Target in Intensive Care Units? Research on Human Tissue, Body Fluids, Neuropsychological Assessment and Brain Imaging
Brief Title: The Gut Microbiome - Source of Sepsis and Novel Target in Intensive Care Units?
Acronym: MS-ICU
Status: Recruiting | Type: Observational
Sponsor: Jena University Hospital (Other)
Collaborators: Friedrich Schiller University of Jena (Unknown)
Responsible Party: Principal Investigator, Johannes Ehler, Principal Investigator, Jena University Hospital
Other Study IDs: 2024-3429-BO
Record Dates: First submitted 2024-12-23; First posted 2024-12-27 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Critical Illness; Intensive Care Unit Delirium; Neurocognitive Deficit; Microbiome,immune Function, Critically Ill; Infection in ICU; Sepsis
Keywords: sepsis; broad-spectrum antibiotics; stool; neuropsychological assessment; delirium; neurocognitive impairment; microbiome
MeSH Terms: conditions — Critical Illness; Sepsis; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and stool samples as well as rectal swaps.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- ICU patients with antibiotic treatment: ICU patients treated with piperacillin/tazobactam or meropenem
- ICU patients without antibiotic treatment: ICU patients without antibiotic treatment during their ICU stay
- Long-term survivors of critical illness: Long-term survivors at least six months or more after the beginning of critical illness.

SUMMARY:
Here, the investigators propose to study host responses to reduced microbiome complexity driven by treatment with broad spectrum antibiotics in patients with severe infections or sepsis. The proposal aims to combine holistic approaches with emerging experimental technologies to investigate the complex interactions between the gut microbiota and its host and assess the impact of specific bacterial communities on longevity and stress responses. A strong focus of this study will also be placed on microbiome dysbiosis and secondary impacts on short- and long-term brain dysfunction using clinical, laboratory and imaging procedures.

DETAILED DESCRIPTION:
Prospective observational study to obtain faeces, rectal swabs, and plasma samples from critically ill patients with and without broad spectrum antimicrobial therapy as well as from long-term survivors after sepsis. Furthermore, clinical, neuropsychological and neuroimaging data will be collected to assess short- and long-term brain dysfunction.

Furthermore it will be to correlate metagenomic and metabolomic data analysis from stool and blood samples of ICU patients with clinical outcomes (including the trajectory of neuro-cognitive deficits) and stress-related parameters.

Additionally, the study aims to identify if microbiome dysbiosis is connected to short- and long-term brain dysfunction and to assess which microbiome metabolic products influence brain dysfunction.

Moreover, the investigators aim to explore immune cell diversity through single cell whole transcriptome analysis in order to establish new hypotheses on specific bacteria species and metabolites to affect the immune cell type composition of patients (single cell immuno-profiling) and integrate single cell RNA sequencing with clinical symptoms in critically ill patients.

Finally, the question is addressed whether there are differences between blood cell composition and activation between younger and older patients with and without sepsis.

In this regard, blood- and stool samples will be taken from participants at five time points as follows: three time points during ICU treatment respectively (at study inclusion day 1, day 7 and day 14) and as well as two follow-up surveys (3 and 6 months after inclusion). Brain dysfunction will be assed by daily delirium screening tests (CAM-ICU and ICDSC) and at the time of discharge from hospital by MoCa and Mini Mental Status Examination. At the follow-up survey functional MRI as well as neuropsychological measures will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* One of the following criteria

  1. Critically ill patients treated with meropenem or piperacillin/tazobactam started within the last 72 h
  2. Critically ill patients without systemic antimicrobial therapy within the last 72 hours and an expected ICU length of stay of more than 3 days
  3. Long-term survivors of sepsis, e.g. from pre-existing sepsis cohorts

Exclusion Criteria:

* Inflammatory bowel disease
* Major bowel resection
* Selective decontamination of the oral and digestive tract
* Oral vancomycin therapy
* Immunocompromised patients
* History of chemotherapy during the last 6 months.
* Known travel history to countries to areas of high antimicrobial resistance (>5% according to the report of the European Centre for Disease Prevention and Control and all countries except USA and Canada) within the last 4 weeks
* Acute neurological diseases (e.g., brain ischemia, hemorrhage, meningoencephalitis, tumor)
* Manifest dementia, pre-existing psychiatric diseases (schizophrenia, psychosis)
* Acute brain surgery
* MRI contraindications: pacemakers, hearing aids, neurostimulation, insulin pumps, other potentially ferromagnetic implants, screws, clips, prostheses, metal splinters, etc., pregnancy, claustrophobia, extensive tattoos.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients with and without antibiotic treatment as well as patients with long-term survival after critical illness
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-27 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with brain dysfunction | From enrollment to day 180
  Patients from all three groups will be assessed for microbiome dysbiosis (e.g. shotgun metagenomics), and for brain dysfunction (e.g. CAM-ICU, ICDSC, MoCa, MMST, neuropsychiatric examination, MRI).

SECONDARY OUTCOMES:
Number of patients with survival | From enrollment to the end of study at 180 days
Days on the ICU | From enrollment to the end of study at 180 days
Days on the respirator | From enrollment to the end of study at 180 days
Days with vasopressor support | From enrollment to the end of study at 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Ehler, Priv.-Doz. Dr. med., Principal Investigator — Department of Anesthesiology and Intensive Care Medicine, Jena University Hospital
Locations (1):
- Klinik für Anästhesiologie und Intensivmedizin, Universitätsklinikum Jena, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No